CLINICAL TRIAL: NCT04451044
Title: Distal Evaluation of Functional Performance with Intravascular Sensors to Assess the Narrowing Effect: Guided Physiologic Stenting
Acronym: DEFINE GPS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 190103
Record Dates: First submitted 2020-06-23; First posted 2020-06-30 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Coronary Artery Disease; Ischemic Heart Disease
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- physiologically-guided arm (Experimental): Physiologically-guided PCI using the Philips SyncVision system for determining the PCI strategy
  Interventions: Device: Philips SyncVision system with Philips pressure wires
- angiographically-guided arm (Active Comparator): Standard of care angiographically-guided PCI for determining the PCI strategy
  Interventions: Procedure: standard of care angiographically-guided PCI

INTERVENTIONS:
Device: Philips SyncVision system with Philips pressure wires — Intent to use physiologically-guided PCI using the Philips SyncVision system for determining the PCI strategy
  Arms: physiologically-guided arm
Procedure: standard of care angiographically-guided PCI — Intent to use PCI standard of care angiographically-guided PCI for determining the PCI strategy
  Arms: angiographically-guided arm

SUMMARY:
Multi-center, prospective, randomized controlled study comparing PCI guided by angiography versus iFR Co-Registration using commercially available Philips pressure guidewires and the SyncVision co-registration system, employing an adaptive design study for interim sample size re-estimation.

DETAILED DESCRIPTION:
DEFINE GPS Substudy: Characterization of Intermediate Lesions (ChIL) will enroll approximately 350 patients at up to 20 sites. This multi-center, prospective, registry will enroll patients consented to be randomized into the DEFINE GPS study but ultimately screen fail. Baseline patient medical and demographic data will be collected along with angiographic and functional data from vessels with intermediate disease deferred from revascularization and will be used to establish a body of imaging data that can be used to validate new image-based physiology applications.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult men and women (local age of consent) who present with stable or unstable angina, or NSTEMI.
* 2. Undergoing cardiac catheterization with planned PCI or possible ad hoc PCI
* 3. Following angiography, PCI is indicated in at least one coronary artery* on the basis of one or more of the following:

  1. Presenting with NSTE-ACS (unstable angina with ECG changes or cardiac enzyme-positive NSTEMI) with an identified culprit lesion with DS ≥50%;
  2. One or more angiographic stenoses present with ≥80% stenosis severity by visual estimation;
  3. One or more angiographic stenoses present with ≥50% to <80% stenosis severity by visual estimation and an abnormal non-invasive stress test in the distribution of the lesion(s) within the past 60 days;
  4. One or more angiographic stenoses are present with ≥50% to <80% stenosis severity by visual estimation and a spot iFR measure ≤0.89 or FFR≤0.80 for borderline iFR..
* 4 Subject is willing to comply with all scheduled visits and tests and has provided informed written consent

Exclusion Criteria:

* 1. STEMI within 30 days
* 2. PCI within the prior 12 months, or any PCI planned after the study procedure (other than planned staged procedures of randomized vessels which are allowed)
* 3. Prior CABG anytime
* 4. Silent ischemia only (i.e. no cardiac symptoms related to coronary artery disease) within the prior 4 weeks
* 5. Documented prior iFR pullback performed in any coronary artery including during the qualifying diagnostic angiogram
* 6. Any vessel with in-stent restenosis (ISR) requiring treatment
* 7. Cardiogenic shock defined as systolic blood pressure <90 mmHg for >20 minutes not responding to fluid resuscitation, or need for inotropic, pressor, or device-based hemodynamic support
* 8. Presence of unstable ventricular arrhythmias
* 9. Heart rate > 110, including uncontrolled atrial fibrillation (AF)
* 10. Decompensated congestive heart failure (NYHA Class IV or Killip Class III or IV)
* 11. Chronic total occlusion (CTO) of a target vessel (exception: a CTO may be present in a non-target vessel if it is supplying non-viable myocardium and there is no intent to open the CTO during the index or later procedure)
* 12. Coronary anatomy not amenable to pressure wire manipulation due to extreme tortuosity or complexity such that it is unlikely that a pressure wire could be passed to the distal third of the three major epicardial coronary arteries
* 13. Any angiographic giant thrombus (i.e., thrombus length > 3x RVD at lesion)
* 14. Any target vessel with < TIMI III flow
* 15. Any target lesion with a reference vessel diameter (RVD) less than 2.25mm except for within the side branch of a bifurcation lesion
* 16. Any non-target lesion with a reference vessel diameter (RVD) greater than 2.00mm that contains an ≥80% stenosis and is not intended for treatment with PCI (other than a CTO supplying non-viable myocardium - see exclusion #11)
* 17. Known severe aortic or mitral valve stenosis/insufficiency
* 18. Known non-cardiovascular comorbidity resulting in lifespan <24 months
* 19. Known left ventricular ejection fraction ≤30%
* 20. Estimated creatinine clearance (MDRD formula) <30 mL/min/1.73m2 or on dialysis
* 21. Any cardiac or non-cardiac surgical procedure planned within 12 months after enrollment, or any procedure planned within 6 months after enrollment that would necessitate discontinuation of dual antiplatelet therapy
* 22. Known pregnancy or planning to become pregnant (women of child-bearing potential must have a negative pregnancy test within 1 week of enrollment)
* 23. Participating in another investigational drug or device study that has not reached its primary endpoint
* 24. Any condition such as dementia or substance abuse that may impair the patient's ability to comply with all study procedures, including medication compliance and follow-up visits
* 25. Patient is a member of a vulnerable population who, in the judgment of the investigator, is unable to give Informed Consent for reasons of incapacity, immaturity, adverse personal circumstances or lack of autonomy. This may include individuals with mental disability, persons in nursing homes, children, impoverished persons, persons in emergency situations, homeless persons, nomads, refugees, and those permanently incapable of giving informed consent. Vulnerable populations also include university students, subordinate hospital and laboratory personnel, employees of the Sponsor, members of the armed forces, and persons kept in detention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3212 (Estimated)
Dates: Start 2021-06-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events (MACE; composite of cardiac death, target vessel MI (TVMI), or ischemia-driven revascularization) or hospitalization for progressive or unstable angina at 2 years | 2 years

SECONDARY OUTCOMES:
Major Adverse Cardiac Events (MACE; composite of cardiac death, target vessel MI (TVMI), or ischemia-driven revascularization) or hospitalization for progressive or unstable angina | 30 days, 1 year
All-cause, cardiac and non-cardiac mortality | 30 days, 1 year and 2 years
All MI, target vessel MI, non-target vessel MI, procedural MI, non-procedural MI | 30 days, 1 year and 2 years
Ischemia-driven revascularization, including all revascularization, TVR, TLR, non-TLR TVR, and non-TVR | 30 days, 1 year and 2 years
Hospitalization for progressive or unstable ischemia | 30 days, 1 year and 2 years
Stent thrombosis (definite, probable and definite/probable) | 30 days, 1 year and 2 years
Angina-related Quality of Life | 30 days, 1 year and 2 years
  Change from baseline in the Seattle Angina Questionnaire (SAQ-7) summary score
Resource utilization | 30 days, 1 year and 2 years
  The [US-based] cost of all health care resources associated with the index procedure and pre-specified event costs throughout the two-year follow up period
Cost effectiveness | 30 days, 1 year and 2 years
  Cost per quality-adjusted life years gained

CONTACTS AND LOCATIONS:
Overall Officials: Allen Jeremias, MD MSC FACC FSCAI, Principal Investigator — Saint Francis Hospital; Gregg W Stone, MD, Study Chair — The Zena and Michael A. Wiener Cardiovascular Institute, Icahn School of Medicine at Mount Sinai
Locations (84):
- United States (40):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Pima Heart & Vascular, Tucson, Arizona
  - Central Arkansas Veterans Healthcare System (CAVHS), Little Rock, Arkansas
  - Glendale Adventist, Glendale, California
  - Colorado Heart and Vascular, Lakewood, Colorado
  - Yale University, New Haven, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Memorial Healthcare, Hollywood, Florida
  - Tampa Cardiovascular Innovations and Research, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Straub Medical Center, Honolulu, Hawaii
  - Carle Foundation Hospital, Urbana, Illinois
  - Community Healthcare System, Munster, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Mass General, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Metro Cardiology Consultants, Coon Rapids, Minnesota
  - Fairview Health Services, Edina, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Gates Vascular Institute, Buffalo, New York
  - Northwell Health, Lake Success, New York
  - Columbia University Medical Center, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - NC Heart and Vascular Research, LLC, Raleigh, North Carolina
  - Summa Health System, Akron, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Jefferson Einstein Medical Center, Philadelphia, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - North Central Heart, Sioux Falls, South Dakota
  - Centennial Medical Center, Nashville, Tennessee
  - Ascension Saint Thomas, Nashville, Tennessee
  - Baylor Scott & White, The Heart Hospital Plano, Plano, Texas
  - Sentara Health, Norfolk, Virginia
  - Carilion Clinic, Roanoke, Virginia
  - Gundersen Health, La Crosse, Wisconsin
- Australia (6):
  - Gosford Hospital, Gosford, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - Lake Macquarie Private Hospital, Gateshead
  - The Alfred Hospital, Melbourne
- Akademisches Lehrkrankenhaus Feldkirch, Feldkirch, Austria
- Canada (5):
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Montreal Heart Institute, Montreal, Quebec
  - William Osler Health-Brampton Civic Hospital, Brampton
  - Hopital du Sacre-Coeur de Montreal, Montreal
  - St. Michael's Hospital, Toronto
- Aarhus University Hospital, Aarhus, Denmark
- France (2):
  - CHU Lille, Institut Coeur Poumon, Lille
  - CHU Nimes Caremeau, Nîmes
- Germany (4):
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Erlangen University Hospital, Erlangen
  - University Hospital Essen, Essen
  - Universitsklinik Freiburg, Freiburg im Breisgau
- Israel (2):
  - Hillel Yaffe Medical Center, Hadera
  - Shamir Medical Center, Tel Aviv
- Careggi University Hospital, Florence, Italy
- Hospital General Querétaro, Querétaro, Mexico
- Netherlands (5):
  - Albert Schweitzer Ziekenhuis / Hartcentum Dordrecht- Gorinchem, Dordrecht
  - Medisch Spectrum Twente, Enschede
  - Medisch Centrum Leeuwarden, Leeuwarden
  - St Antonius Hospital Nieuwegein, Nieuwegein
  - Radboud University Med Ctr, Nijmegen
- Medical University of Warsaw, Warsaw, Poland
- Hospital Prof. Doutour Fernando Foneseca, Amadora, Portugal
- South Korea (3):
  - Sejong General Hospital, Bucheon-si
  - Keimyung University Dongsan Medical Center, Daegu
  - Seoul National University Hospital, Seoul
- Spain (4):
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario de Leon, León
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Marqués de Valdecillas, Santander
- Sweden (2):
  - Skane University Hospital, Lund
  - Örebro University Hospital, Örebro
- Geneva University Hospital, Geneva, Switzerland
- United Kingdom (4):
  - University Hospital Southampton, Southampton, Hampshire
  - University Hospital of Wales, Cardiff, Wales
  - Royal Bournemouth Hospital, Bournemouth
  - Imperial College Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: No